CLINICAL TRIAL: NCT01307631
Title: A Phase II, 2-Stage, 2-Arm PIK3CA Mutation Stratified Trial of MK-2206 in Recurrent or Advanced Endometrial Cancer
Brief Title: Akt Inhibitor MK2206 in Treating Patients With Recurrent or Advanced Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00521; NCI-2013-00521 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10.258; 10-258 (Other: Dana-Farber Cancer Institute); 8760 (Other: CTEP); P30CA006516 (NIH); U01CA062490 (NIH); UM1CA186709 (NIH); NCT01312753 (obsolete NCT alias)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Adenosquamous Carcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Recurrent Uterine Corpus Carcinoma
MeSH Terms: interventions — MK 2206

ARMS (1):
- Treatment (Akt inhibitor MK2206 (Experimental): Patients receive Akt inhibitor MK2206 PO once weekly. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well Akt inhibitor MK2206 works in treating patients with recurrent or advanced endometrial cancer. Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of MK-2206 (Akt inhibitor MK2206) in patients with recurrent or persistent endometrial cancer classified by phosphoinositide-3-kinase catalytic alpha (PIK3CA) mutation. Activity will be ascertained by the proportion of patients who survive progression-free for at least 6 months after initiating therapy or who have objective tumor response.

II. To evaluate the efficacy of MK2206 in patients with serous tumors using a composite endpoint of complete and partial response by Response Evaluation Criteria In Solid Tumors (RECIST) and progression-free interval of 6 months or longer.

SECONDARY OBJECTIVES:

I. To determine the duration of progression-free survival and overall survival. II. To determine the nature and degree of toxicity of MK-2206 as assessed by version 4 of the National Cancer Institute (NCI) Common Terminology Criteria For Adverse Events (CTCAE) in these cohorts of patients.

III. To explore the associations between select biomarkers and response to MK-2206 such as progression-free survival, objective tumor response, and overall survival as well as patient characteristics such as histological cell type.

IV. To explore the development of feed-back loop activation (post-treatment biopsy biomarker analysis) and target inhibition using MK-2206 via analysis of pre-treatment and post-treatment biopsies in select patients enrolled in the trial.

V. To determine the duration of progression-free and overall survival, following initiation of therapy with MK-2206.

VI. To determine the toxicities of MK-2206, as assessed with the revised NCI CTCAE version 4.

VII. To explore the association between select biomarkers and response to MK-2206 such as progression-free survival, objective tumor response.

OUTLINE:

Patients receive Akt inhibitor MK2206 orally (PO) once weekly. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed recurrent or persistent high grade endometrial carcinoma with a serous component, which is refractory to curative therapy or established treatments; histologic confirmation of the original primary tumor is required
* All patients must have measurable disease as defined by RECIST 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have had one prior chemotherapeutic regimen for management of endometrial carcinoma initial treatment may include chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy; chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen
* Patients are allowed to receive, but are not required to receive, one additional prior treatment regimen (including a single chemotherapeutic, a combination of chemotherapeutics, or an anti-angiogenic drug such as bevacizumab) for management of their recurrent or persistent disease; prior hormonal therapy is allowed and does not count towards this prior regimen
* Patients must have NOT received any class of drugs targeted to the PI3K pathway (such has PI3K inhibitors or mTOR inhibitors) for management of recurrent or persistent disease
* Life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits or creatinine clearance >= 60 mL/min/1.73 m^2 for subjects with creatinine levels about institutional normal
* Hemoglobin A1c (HgA1c) =< 7.5% and fasting blood glucose less than 130mg/dL
* Availability of a formalin fixed paraffin embedded (FFPE) block of cancer tissue from the original or most recent biopsy for mutational analysis
* Women of childbearing potential must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a patient become pregnant or suspect she is pregnant while she is participating in this study, she should inform the treating physician immediately
* Toxicities of prior therapy (excepting alopecia) should be resolved to =< grade 1 per the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4
* MK-2206 is an oral medication; patients must be able to tolerate oral medications and not have gastrointestinal illnesses that would preclude absorption of MK-2206
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered to =< grade 1 (excepting alopecia) from adverse events (as per the revised NCI CTCAE version 4) due to agents administered more than 3 weeks earlier
* Participants may not be receiving any other study agents
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; should patients develop brain metastases while on trial and have clinical benefit from MK-2206 otherwise, patients may continue on drug after clinical management of the brain metastases with the permission of the principal investigator. MK-2206 should be restarted between 3 and 6 weeks after the last radiation treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206
* Patients requiring any medications or substances that are strong inhibitors or inducers of CYP 450 3A4 are ineligible
* Preclinical studies demonstrated the potential of MK-2206 for induction of hyperglycemia in all preclinical species tested; patients with diabetes or in risk for hyperglycemia should not be excluded from trials with MK-2206, but the hyperglycemia should be well controlled on oral agents before the patient enters the trial. HgbA1c > 7.5% or fasting glucose greater than 130mg/dL will exclude patients from entry on study; patients requiring insulin for control of their hyperglycemia are excluded from entry on this study
* Preclinical studies indicated transient changes in QTc interval during MK-2206 treatment; prolongation of QTc interval is potentially a safety concern while on MK-2206 therapy; cardiovascular: baseline QTcF > 450 msec (male) or QTcF > 470 msec (female) will exclude patients from entry on study
* Due to a high incidence of bradycardia by Holter monitor, preexisting bundle branch block or baseline bradycardia due to cardiac disease will exclude patients from treatment with MK-2206
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; mother with MK-2206 breastfeeding should be discontinued if the mother is treated with MK-2206; these potential risks may also apply to other agents used in this study
* MK-2206 is an oral medication; patients who are unable to tolerate oral medication are not eligible; patients with signs and symptoms of bowel obstruction or with uncontrolled, persistent diarrhea will be excluded
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: breast cancer in situ, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin
* Human immunodeficiency virus (HIV)-positive individuals on combination antiretroviral therapy are ineligible
* Patients may not use natural herbal products or other "folk remedies" while participating in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2015-09-18 (Actual); Study Completion 2015-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Konstantinopoulos, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Myers AP, Konstantinopoulos PA, Barry WT, Luo W, Broaddus RR, Makker V, Drapkin R, Liu J, Doyle A, Horowitz NS, Meric-Bernstam F, Birrer M, Aghajanian C, Coleman RL, Mills GB, Cantley LC, Matulonis UA, Westin SN. Phase II, 2-stage, 2-arm, PIK3CA mutation stratified trial of MK-2206 in recurrent endometrial cancer. Int J Cancer. 2020 Jul 15;147(2):413-422. doi: 10.1002/ijc.32783. Epub 2019 Dec 13. PMID 31714586

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Akt Inhibitor MK2206) PIK3CA Mutation: Patients with PIK3CA mutation receive Akt inhibitor MK2206 PO once weekly. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Akt Inhibitor MK2206: Given PO
  Laboratory Biomarker Analysis: Correlative studies
- Treatment (Akt Inhibitor MK2206) Wild Type: Patients with wild type receive Akt inhibitor MK2206 PO once weekly. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Akt Inhibitor MK2206: Given PO
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Akt Inhibitor MK2206) PIK3CA Mutation | Treatment (Akt Inhibitor MK2206) Wild Type
Started | 9 | 28
Completed | 9 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Akt Inhibitor MK2206
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 56 [39 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response According to RECIST
Description: Activity will be ascertained by the proportion of patients who survive progression-free for at least 6 months after initiating therapy or who have objective tumor response. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to < 10 mm; Partial Response (PR), at least 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 6 months
Population: Number of patients who had an objective response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Akt Inhibitor MK2206
Number analyzed (Participants) | 37
Participants | 2

2. Primary Outcome: Progression-free Survival According to RECIST
Description: as for outcome 1
Time Frame: From start of treatment to time of objective disease progression, assessed up to 6 months
Population: Number of patients who had a PFS > 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Akt Inhibitor MK2206
Number analyzed (Participants) | 37
Participants | 4

3. Secondary Outcome: Duration of Overall Survival
Description: Estimated by using Kaplan-Meier analysis.
Time Frame: Up to 3 years
Population: Overall survival of all patients on study.
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Akt Inhibitor MK2206
Number analyzed (Participants) | 37
months | 8 [0 to 12]

4. Secondary Outcome: Duration of Progression-free Survival
Description: Estimated by using Kaplan-Meier analysis.
Time Frame: Up to 3 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Akt Inhibitor MK2206) PIK3CA Mutation | Treatment (Akt Inhibitor MK2206) Wild Type
Number analyzed (Participants) | 9 | 28
months | 1.6 [0 to 1.6] | 1.8 [0 to 1.8]

5. Other Pre Specified Outcome: Association Between Select Biomarkers and Response to Akt Inhibitor MK2206 Such as Progression-free Survival and Objective Tumor Response, Assessed by Immunohistochemistry (IHC)
Time Frame: Up to 3 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Incidence of Adverse Events as Assessed by NCI CTCAE Version 4.0 [Time Frame: Up to 3 Years] [Designated as Safety Issue: Yes]
Description: Data is reported in the Adverse Event table.
Time Frame: 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the treatment start of the patient to 30 days after the patient has come off treatment.
Arm/Group | Treatment (Akt Inhibitor MK2206
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 14/37
Other Adverse Events (participants affected / at risk) | 15/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206 (N=37)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Hyperglycemia (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Thromboembolic event (Blood and lymphatic system disorders) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206 (N=37)
abdominal pain (Gastrointestinal disorders) | 4 (5)
Acute kdiney injury (Renal and urinary disorders) | 2 (2)
edema limbs (General disorders) | 5 (5)
anorexia (Metabolism and nutrition disorders) | 3 (3)
creatinine decreased (Investigations) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 6 (6)
fatigue (General disorders) | 11 (13)
constipation (Gastrointestinal disorders) | 5 (6)
diarrhea (Gastrointestinal disorders) | 6 (8)
urinary tract infections (Infections and infestations) | 2 (2)
hyponatremia (Metabolism and nutrition disorders) | 1 (2)
skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
pelvic pain (Reproductive system and breast disorders) | 2 (2)
vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 5 (5)
anxiety (Psychiatric disorders) | 1 (1)
hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
insomnia (Psychiatric disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 2 (5)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 3 (3)
weight loss (Investigations) | 1 (1)
hot flashes (Vascular disorders) | 1 (1)
bruising (Injury, poisoning and procedural complications) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
non-cardiac chest pain (General disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
urinary frequency (Renal and urinary disorders) | 1 (2)
hematuria (Renal and urinary disorders) | 1 (1)
creatinine increased (Investigations) | 1 (2)
bone pain (Musculoskeletal and connective tissue disorders) | 2 (4)
ataxia (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less